CLINICAL TRIAL: NCT02669550
Title: A Comparison of Disposcope Endoscope and Fiberoptic Bronchoscope During Awake Orotracheal Intubation in Obese Patients With Anticipated Difficult Airway : A Prospective, Randomised and Controlled Clinical Trial
Brief Title: Comparison of Disposcope Endoscope and Fiberoptic Bronchoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 0001
Record Dates: First submitted 2015-11-22; First posted 2016-02-01 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2016-01

CONDITIONS: Therapeutic Procedural Complication
Keywords: Fiberoptic bronchoscope; Disposcope endoscope; Awake orotracheal intubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fiberoptic bronchoscope (Experimental): In case of FOB, the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Interventions: Device: Fiberoptic bronchoscope
- Disposcope endoscope (Experimental): In the DE group, the operator gripped the chin and lower incisors of patients with the fingers and thumb to open the mouth adequately wide and grasped the wire body, which was enclosed within the endotracheal tube, by the other hand and held it parallel to,then inserted into oral cavity
  Interventions: Device: Disposcope endoscope

INTERVENTIONS:
Device: Fiberoptic bronchoscope — In case of FOB, the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Arms: Fiberoptic bronchoscope
Device: Disposcope endoscope — In the DE group, the operator gripped the chin and lower incisors of patients with the fingers and thumb to open the mouth adequately wide and grasped the wire body, which was enclosed within the endotracheal tube, by the other hand and held it parallel to,then inserted into oral cavity
  Arms: Disposcope endoscope

SUMMARY:
The fiberoptic bronchoscope (FOB) has been the preferred instrument for many years in the management of difficult tracheal intubation, and it is considered as a gold standard. The disposcope endoscope (DE) is a medical device for endotracheal intubation used in clinical practice recently.This study compares FOB and DE for awake orotracheal intubation in obese patients with anticipated difficult airway.

DETAILED DESCRIPTION:
Forty obese patients with anticipated difficult airways were randomised to undergo awake orotracheal intubation by FOB(group F) or DE(group D) after conscious sedation. The conditions of orotracheal intubation, the time needed to view the vocal cords and to complete the orotracheal intubation, the hemodynamic changes and the adverse events including bradycardia, respiratory depression during orotracheal intubation, throat pain, hoarseness and memory after surgery were recorded. The ease of view the vocal cords and passing the tracheal tube through the glottis were also evaluated by using a visual analogue scale (VAS) by operator.

ELIGIBILITY:
Inclusion Criteria:

* ASA classifications of I-II, modified Mallampati classification of 3 or 4, requiring general anesthesia were included.

Exclusion Criteria:

* Exclusion criteria included age younger than 18 yr,
* ASA class IV or V,
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intubation Time | 36 months

SECONDARY OUTCOMES:
Occurrence of throat pain measured by VAS | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, PHD, Study Director — The First Hospital of Qinhuangdao

IPD SHARING:
Plan to Share IPD: Yes